CLINICAL TRIAL: NCT04487808
Title: Cardiometabolic Effects of Including Pecans as a Snack in Dietary Patterns That Vary in Diet Quality: a Randomized, Controlled Feeding, Crossover Study
Brief Title: Diet Quality, Pecans, and Cardiometabolic Health
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study did not enroll any subjects. It was never started because of the Covid pandemic.
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Pecan
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Average American Diet (Active Comparator): Diet representative of average American intake in terms of diet quality measured by the Healthy Eating Index-2015.
  Interventions: Other: Average American Diet devoid of nuts
- Average American Diet + Pecans (Active Comparator): Diet that approximates average American intake in terms of diet quality measured by the Healthy Eating Index-2015, but includes 2 oz./day of pecans.
  Interventions: Drug: Pecan
- Healthy Diet + Pecans (Active Comparator): High diet quality, measured by Healthy Index-2015 score >95, and includes 2 oz./day of pecans.
  Interventions: Drug: Pecan

INTERVENTIONS:
Drug: Pecan — Unsalted raw pecans incorporated in snack and meal recipes as part of a dietary pattern
  Arms: Average American Diet + Pecans; Healthy Diet + Pecans
Other: Average American Diet devoid of nuts — Diet mimicking usual American intake
  Arms: Average American Diet

SUMMARY:
A three-period, randomized, crossover controlled feeding trial will be conducted to examine the effect of including 2 oz./day of pecans, as a snack, in a diet representative of average American intake, compared to a diet representative of average American intake devoid of nuts, and a healthy dietary pattern including 2 oz./day of pecans on markers of peripheral vascular health, lipids and lipoproteins, blood pressure, and glycemic control.

DETAILED DESCRIPTION:
Participants will be randomized to each diet for 4-weeks with a minimum 2-week break between the diet periods. All caloric foods and beverages will be provided. Outcome assessments will be done at baseline and the end of each diet period.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25 and ≤40 kg/m2
* ≥ 1 criterion for metabolic syndrome (i.e. waist circumference ≥ 94 cm men or ≥80 cm women; triglycerides ≥150 mg/dL; HDL ≤ 40 mg/dL men or ≤50 mg/dL women; systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg; fasting plasma glucose ≥100 mg/dL) at screening.
* non-smoking

Exclusion Criteria:

* Current tobacco use or use within the previous 6 months
* Diagnosed diabetes or fasting glucose levels > 126 mg/dL at screening
* Systolic blood pressure >160 mm Hg or diastolic blood pressure > 100 mm Hg at screening.
* Use of anti-hypertensive, lipid lowering, glucose lowering drugs, steroids, or antibiotics in the previous month
* History of a cardiovascular event (heart attack, revascularization, stroke), or heart failure, liver, kidney, autoimmune diseases or inflammatory conditions such as gastrointestinal disorders or rheumatoid arthritis
* Use of supplements and botanicals known to affect study outcomes (e.g. psyllium, fish oil, soy lecithin, and phytoestrogens) and not willing to cease for the duration of the study
* Pregnancy, lactation or planning to become pregnant
* Consumption of >14 alcoholic drinks/week
* Intolerance/allergy/sensitivity to foods included in the study menus

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Flow mediated dilation | 4 weeks
  Measured by brachial ultrasound and expressed as percent artery dilation

SECONDARY OUTCOMES:
LDL-cholesterol concentration | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL
HDL-cholesterol concentrations | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL
Triglycerides | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL
LDL lipoprotein subclasses | 4 weeks
  Assessed from fasting blood draw expressed in nmol/L
HDL lipoprotein subclasses | 4 weeks
  Assessed from fasting blood draw expressed in umol/L
Peripheral systolic and diastolic blood pressure | 4 weeks
  Blood pressure measured assessed using a SphymoCor Ecel (Atcor Medical)
Central systolic and diastolic blood pressure | 4 weeks
  Blood pressure measured assessed using a SphymoCor Ecel (Atcor Medical).
Carotid-femoral pulse wave velocity | 4 weeks
  A measure of arterial stiffness assessed using a SphymoCor Ecel (Atcor Medical). Expressed in meters/second.
Augmentation Index | 4 weeks
  A measure of arterial stiffness assessed using a SphymoCor Ecel (Atcor Medical). Expressed as a percentage. A higher percentage value is indicative of greater arterial stiffness.
Fasting plasma glucose concentration | 4 weeks
  Fasting blood glucose assessed by blood draw and expressed in mg/dL
Serum insulin concentration | 4 weeks
  Fasting serum insulin levels assessed by blood draw and expressed in micro IU/mL

OTHER OUTCOMES:
Change in the composition of the gut microbiota | 4 weeks
  Abundance measured using 16 s rRNA sequencing

IPD SHARING:
Plan to Share IPD: No